CLINICAL TRIAL: NCT02243449
Title: Screening Elderly PatieNts For InclusiOn in a Weaning Trial: The SENIOR Trial
Brief Title: Screening Elderly Patients for Weaning
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SENIOR0000001; ClinicalTrials.gov Identifier: (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2014-04-01; First posted 2014-09-18 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Critically Ill
Keywords: mechanical ventilation; weaning; elderly; critically ill; screening; spontaneous breathing trial; invasive ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Once daily screening (Active Comparator): In the 'once daily screening arm', RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hours of the scheduled screening period. Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol.
  Interventions: Procedure: Once daily screening
- At least twice daily screening (Experimental): In the 'at least twice daily' screening arm patients will be screened at a minimum between approximately 06:00 - 08:00 hours and 13:00 - 15:00 hours daily. If a screening period is missed inadvertently or due to an investigation or intervention (operation/procedure) necessitating absence from the ICU, it may be conducted later on the same day and ideally within 6 hours of the scheduled screening period. Additional screening trials in the 'at least twice daily' screening arm will be permitted at the discretion of the clinical team (RTs and physicians). Regardless of group assignment, if the SBT screening assessment is passed, an SBT will be conducted as per protocol.
  Interventions: Procedure: At least twice daily screening

INTERVENTIONS:
Procedure: Once daily screening — In the 'once daily screening arm', RTs will screen invasively ventilated patients between approximately 06:00 - 08:00 hours daily. To pass the 'readiness to wean screen' and undergo an SBT, specific criteria must be met. The initial SBT will be 30-120 minutes in duration and may be conducted with any one of the following techniques: T-piece, continuous positive airway pressure (CPAP) less than or equal to 5 cm H2O or PS less than or equal to 8 cm H2O with PEEP less than or equal to 5 - 10 cm H2O. Higher levels of PEEP (8-10 cm H2O) will be permitted (and recorded) to allow for clinician discretion in conducting SBTs in specific patients (e.g., obese, chronic obstructive pulmonary disease) and use of different humidification strategies. Each centre will be asked to choose one technique to be used for patients enrolled at their centre.
  Arms: Once daily screening
Procedure: At least twice daily screening — In the 'at least twice daily' screening arm patients will be screened at a minimum between approximately 6:00-8:00 hours and 13:00-15:00 hours daily. To pass the 'readiness to wean screen' and undergo an SBT, specific criteria must be met. The initial SBT will be conducted in the same manner as in the once daily screening arm. The subsequent SBTs will be 30 -120 minutes in duration and may be conducted with any one of the following techniques: T-piece, CPAP < to 5 cm H2 O or PS < 8 cm H2 O with PEEP < 5 - 10 cm H2O. Higher levels of PEEP (8-10 cm H2O) will be permitted (and recorded) to allow for clinician discretion in conducting SBTs in specific patients (e.g., obese, chronic obstructive pulmonary disease) and with the use of different humidification strategies. Each centre will be asked to choose one technique for all patients enrolled at their centre.
  Arms: At least twice daily screening

SUMMARY:
During weaning the work of breathing is transferred from the ventilator back to the patient. Approximately 40% of the time on ventilators is spent weaning. Studies support the use of screening protocols and tests of patient's ability to breathe spontaneously (SBTs) to identify weaning candidates. The investigators work demonstrates that once daily screening is the current standard of care. The conduct of daily ward rounds and once daily screening in ICUs is poorly aligned with the rapidly changing clinical status of critically ill patients. With respiratory therapists (RTs) in Canadian intensive care units (ICUs), a significant opportunity exists to screen patients more often, conduct more SBTs, and reduce the time spent on ventilators and in the ICU. Only one mechanical ventilation trial has focused on the elderly and no trial has evaluated weaning outcomes in the elderly and very elderly which may be influenced by the presence of comorbidities, frailty, malnutrition and treatment limitations.

The investigators propose to conduct a pilot randomized trial in 100 elderly (>/= 65 years) critically ill adults comparing 'once daily' screening to 'at least twice daily' screening in 8 adult ICUs. In the proposed trial, the investigators will (i) evaluate their ability to recruit elderly (>/= 65 years) critically ill patients into a weaning trial and (ii) assess whether protocols can be adhered to similarly between elderly (65 to 80 years) and very elderly (>80 years) trial participants. Moreover, they will also address generalizability issues in the conduct of mechanical ventilation research by evaluating potential biases associated with exclusion criteria and consent between elderly and very elderly patients and obtain preliminary estimates of differences in important clinical outcomes between elderly and very elderly participants.

DETAILED DESCRIPTION:
In the context of a multicentre, pilot trial in 100 elderly (>/= 65 years) critically ill adults comparing two strategies to identify weaning candidates ('once daily' vs. 'at least twice daily' screening) in 8 ICUs across Canada, we propose to assess feasibility metrics that reflect our ability to consent, enroll and recruit elderly and very elderly invasively ventilated patients and evaluate adherence to the study protocols in preparation for launching a large scale screening RCT.

1. Primary Research Question (i) Can we recruit invasively ventilated elderly (age >/= 65 years) critically ill adults into a weaning trial comparing alternative screening strategies?
2. Secondary Research Questions (ii) Can clinicians adhere to the assigned screening protocols in both study arms?
3. Tertiary Research Questions

   (ii) What are the proportions of enrolled elderly and very elderly trial participants? (iii) Are the proportions of consents obtained and declined for trial participation similar between eligible elderly and very elderly trial participants? (iv) What are the rates and reasons for trial exclusion based between eligible elderly and very elderly patients? (v) What effect, in preliminary estimates, do the alternative screening strategies have on clinically important outcomes[e.g., time to first Spontaneous Breathing Trial (SBT) and first successful SBT, time to first extubation and successful extubation, total duration of mechanical ventilation, intensive care unit (ICU) and hospital length of stay, ICU and hospital mortality, use of noninvasive ventilation (NIV) following extubation, complications (self-extubation, tracheostomy, reintubation, proportion requiring prolonged mechanical ventilation) and adverse events] between elderly and very elderly trial participants.
4. Quaternary Research Questions

(i) Can we assess and quantify current practices related to sedation, analgesia an delirium management and mobilization before conducting 'once daily' or 'at least twice daily screening' assessments of weaning readiness with the goal of quantifying factors that may lead to performance bias in the future, planned, large scale weaning trial.

(ii) Can we identify barriers (clinician and institutional) to recruitment into this study? (iii) Can we classify trial participants as requiring (i) simple, (ii) difficult or (iii) prolonged weaning using the 'Task Force on Weaning' definitions.

Hypotheses

We hypothesize that we will achieve our feasibility metrics, specifically, that:

1. We will recruit at least 2 elderly critically ill patients, on average, per month per ICU.
2. Compliance rates will be at least 80% in both study arms and contamination in the once daily screening arm will be < 10%.
3. We expect that we will enroll similar proportions of elderly than very elderly trial participants.
4. We anticipate that the proportion of consents obtained will be similar between eligible elderly and very elderly participants, the rate of declined consents will be higher in very elderly trial participants.
5. We anticipate that rates of exclusion will be greater for very elderly trial participants due to increased prevalence of comorbid illnesses and treatment limitations.
6. We expect that preliminary estimates of the impact of the alternative screening strategies on clinically important outcomes will be similar between elderly and very elderly trial participants.
7. Practices in sedation, analgesia, delirium and mobilization will be recorded at least 80% of the time.
8. We will identify potentially modifiable clinician and institutional barriers to recruitment.
9. Proportions of critically ill adults requiring simple, difficult or prolonged weaning in Canadian ICUs will be similar to those reported in the world literature.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include:

1. elderly (age >/= 65 years) critically ill adults
2. receiving invasive mechanical ventilation for at least 24 hours who can breathe spontaneously on Pressure Support (PS) or trigger breaths on volume or pressure Assist Control (AC), volume or pressure Synchronized Intermittent Mandatory Ventilation (SIMV) ± PS, Pressure Regulated Volume Control (PRVC) or Airway Pressure Release Ventilation (APRV).
3. patients must be receiving </= 70% inspired oxygen
4. and a positive end-expiratory pressure of </= 12 cm H2O (Table 2). .

Exclusion Criteria:

The investigators will exclude patients who have already undergone extubation or an SBT, are unlikely to benefit (e.g. moribund, expected brain death), on automated weaning modes, participating in studies with a weaning protocol, and those who can not be optimized with regard to sedation and mobilization.

Specifically, we will exclude patients:

1. admitted after cardiopulmonary arrest or with brain death or expected brain death,
2. who have evidence of myocardial ischemia in the 24 hour period before enrollment,
3. who have received continuous invasive mechanical ventilation for >/= 2 weeks,
4. who have a tracheostomy in situ at the time of screening,
5. who are receiving sedative infusions for seizures or alcohol withdrawal,
6. who require escalating doses of sedative agents,
7. who are receiving neuromuscular blockers or who have known quadriplegia, paraplegia or 4 limb weakness or paralysis preventing active mobilization (e.g., active range of motion, exercises in bed, sitting at edge of bed, transferring from bed to chair, standing, marching in place, ambulating),
8. who are moribund (e.g., at imminent risk for death) or who have limitations of treatment (e.g., withdrawal of support, do not reintubate order, however, do not resuscitate orders will be permitted),
9. who have profound neurologic deficits (e.g. large intracranial stroke or bleed) or Glasgow Coma Scale (GCS) </= 6,
10. who are using modes that automate SBT conduct,
11. who are current enrolled in a confounding study that includes a weaning protocol,
12. who were previously enrolled in this trial,
13. patients who have already undergone an SBT or
14. patients who have already undergone extubation [planned, unplanned (e.g. self, accidental)] during the same ICU admission.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recruit, on average, 2 elderly invasively ventilated, critically ill patients per ICU per month. | 12 months
  As a feasibility trial, the investigators propose to assess feasibility metrics that reflect their ability to consent, enroll and recruit elderly and very elderly invasively ventilated patients and evaluate adherence to the study protocols in preparation for launching a large scale screening RCT including whether they can recruit invasively ventilated elderly (age >/= 65 years) critically ill adults into a weaning trial comparing the alternative screening strategies.

SECONDARY OUTCOMES:
Adhere to the assigned screening protocols in both study arms. | 12 months
  The investigators will assess whether clinicians can adhere to the assigned screening protocols in both study arms. They will consider compliance rates of at least 80% to be acceptable in both study arms and contamination in the once daily screening arm will be < 10%.

OTHER OUTCOMES:
Proportion of enrolled elderly and very elderly trial participants | 12 months
  Comparison of the proportions of enrolled elderly and very elderly trial participants.
Proportion of consents obtained and declined for trial participation | 12 months
  Compare the proportions of consents obtained and declined for trial participation similar between eligible elderly and very elderly trial participants.
Rates and reasons for trial exclusion | 12 months
  Description of the rates and reasons for trial exclusion based between eligible elderly and very elderly patients.
Effect of the alternative screening strategies on clinically important outcomes (see below) between elderly and very elderly trial participants? | 12 months + 2 months follow up
  Compare, in preliminary estimates, the effect of the alternative screening strategies on clinically important outcomes [time to first SBT, time to first successful SBT, time to first extubation and successful extubation, total duration of mechanical ventilation, ICU and hospital length of stay, ICU and hospital mortality, use of noninvasive ventilation (NIV) after extubation and complications rates [reintubation, self-extubation, tracheostomy, prolonged mechanical ventilation > 7d and > 21 d] and adverse event rates between elderly and very elderly trial participants.

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. A. Burns, MD, FRCPC, Principal Investigator — St. Michael's Hospital (Toronto, Canada)
Locations (8):
- Canada (8):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - St Joseph's Hospital, Hamilton, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hôpital Saint-Luc, Montreal, Quebec
  - Universite Hopitalier de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Burns KEA, Wong JTY, Dodek P, Cook DJ, Lamontagne F, Cohen A, Mehta S, Kho ME, Hebert PC, Aslanian P, Friedrich JO, Brochard L, Rizvi L, Hand L, Meade MO, Amaral AC, Seely AJ; Canadian Critical Care Trials Group. Frequency of Screening for Weaning From Mechanical Ventilation: Two Contemporaneous Proof-of-Principle Randomized Controlled Trials. Crit Care Med. 2019 Jun;47(6):817-825. doi: 10.1097/CCM.0000000000003722. PMID 30920411